CLINICAL TRIAL: NCT02922933
Title: An Open-Label, 3-Part, 2-Period Study to Examine the Effect of Omeprazole (Part 1), Famotidine (Part 2), and of an Acidic Beverage (Part 3) on the Single-Dose Pharmacokinetics of Entinostat in Healthy Adult Subjects
Brief Title: A Study to Examine the Effect of Omeprazole, Famotidine, and an Acidic Beverage on the Pharmacokinetics of Entinostat in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SNDX-275-0150
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Volunteers; Healthy Volunteers; Human Volunteers; Normal Volunteers
Keywords: entinostat; Histone Deacetylase Inhibitor; HDAC
MeSH Terms: interventions — entinostat; Omeprazole; omeprazole, sodium bicarbonate drug combination; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omeprazole (Active Comparator): Treatment A: 5mg entinostat on Day 1
  Treatment B: 20mg omeprazole for 5 days with 5mg entinostat on Day 1
  Interventions: Drug: entinostat; Dietary Supplement: Omeprazole
- Famotidine (Active Comparator): Treatment C: 5mg entinostat on Day 1
  Treatment D: 20mg famotidine on Days -1 and 1 with 5mg entinostat on Day 1
  Interventions: Drug: entinostat; Dietary Supplement: Famotidine
- Acidic Beverage (Active Comparator): Treatment E: 20mg omeprazole for 5 days with 5mg entinostat on Day 1 taken with water
  Treatment F: 20mg omeprazole for 5 days with 5mg entinostat on Day 1 taken with an acidic beverage
  Interventions: Drug: entinostat; Dietary Supplement: Omeprazole

INTERVENTIONS:
Drug: entinostat — HDAC (histone deacetylase inhibitor)
  Other Names: SNDX-275; MS-275
Dietary Supplement: Omeprazole — Proton pump inhibitor
  Other Names: Prilosec; Zegerid
  Arms: Acidic Beverage; Omeprazole
Dietary Supplement: Famotidine — Histamine-2 blocker
  Other Names: Pepcid
  Arms: Famotidine

SUMMARY:
The purpose of this study is therefore to evaluate the effect of concomitant drugs through an increase of intra-gastric pH levels on the bioavailability of entinostat.

The primary objectives of this study are to evaluate the effect of multiple doses of omeprazole, famotidine, and the effect of an acidic beverage in combination with omeprazole on the single-dose PK profile of entinostat.

The secondary objectives are to evaluate the safety and tolerability of a single dose of entinostat when administered with multiple doses of omeprazole, famotidine, and when administered with an acidic beverage in combination with omeprazole.

DETAILED DESCRIPTION:
This is a 3-part study. A total of 204 subjects will be dosed in this study if Parts 2 and 3 are conducted.

In Part 1, in Period 1, a single dose of entinostat will be administered. In Period 2, multiple doses of omeprazole will be administered for 5 days with a single dose of entinostat co-administered. If preliminary results in Period 2 of Part 1 indicate that omeprazole exhibits clinically significant drug-drug interaction (DDI) with entinostat, then Parts 2 and 3 will be conducted. If no DDI interaction is concluded between entinostat and omeprazole in Part 1, then neither Part 2 nor 3 will be conducted.

Part 2 will investigate the effect of multiple doses of famotidine administration on entinostat PK. In Period 1, a single dose of entinostat will be administered. In Period 2, oral doses of famotidine with a single dose of entinostat co-administered.

Part 3 will evaluate the effect of an acidic beverage co-administered with entinostat in subjects with increased gastric pH due to omeprazole treatment. In Period 1, multiple oral doses of omeprazole will be administered with a single dose of entinostat co-administered with water. In Period 2, multiple doses of omeprazole will be administered with a single dose of entinostat co-administered with an acidic beverage.

In all parts, PK samples will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 19-55 years of age at screening.
* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to first dose and throughout the study.
* Body mass index of ≥ 18.5 at screening.
* Medically healthy with no significant medical history, physical examination, laboratory values, vital signs, or ECGs. Liver function tests and serum bilirubin must be ≤ the upper limit of normal. Platelets, hemoglobin, and hematocrit must be > the lower limit of normal at screening.
* Females of non-childbearing potential must have undergone sterilization procedures as noted in the protocol at least 6 months prior to first dose.
* Non-vasectomized male subjects must agree to use a condom with spermicide or abstain from sexual intercourse during the study and until 90 days beyond dose of study drug.
* Male subjects must agree not to donate sperm from the first dose and until 90 days beyond dose of study drug.
* For Part 3 only, must be able to consume approximately 240 mL of a non-diet cola beverage within approximately 3 minutes.
* Understands the study procedures in the informed consent form and be willing and able to comply with the protocol.

Exclusion Criteria:

* Mentally or legally incapacitated or has significant emotional problems at screening or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* History of illness that might confound the results of the study or poses an additional risk to the subject by their participation in the study in the opinion of the PI or designee.
* History of presence of alcoholism or drug abuse within the past 2 years prior to dose.
* History or presence of hypersensitivity or idiosyncratic reaction to entinostat, omeprazole, famotidine, or Coca-Cola(r) Classic.
* History or presence of clinically significant cancer, cardiovascular disorders, acute or chronic gastrointestinal conditions in the opinion of the PI.
* Females of childbearing potential.
* Females with a positive pregnancy test or lactating.
* Positive H. pylori breath test at screening for Parts 1 and .
* Positive urine drug or alcohol results are screening or each check-in.
* Positive urine cotinine at screening.
* Positive results are screening for HIV, hepatitis B surface antigen, or hepatitis C virus
* Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
* Seated heart rate lower than 40 bpm or higher than 99 bpm at screening.
* QTcB interval (correction value of the interval between the Q and T waves on the ECG tracing using the Bazett Correction Formula) > 460 msec for males or > 480 msec for females or has ECG findings deemed abnormal by the PI or designee.
* Estimated creatinine clearance < 90 mL/min at screening.
* Unable to refrain from or anticipates the use of any prescription or non-prescription medications and any drugs known to be significant inhibitors or CYP (Cytochromes 450) enzymes and/or P-gp.
* Has been on a diet incompatible with the on-study diet within 28 days prior to dose and throughout the study in the opinion of the PI or designee.
* Donation of blood or significant blood loss within 56 days prior to dose.
* Plasma donation within 7 days prior to dose.
* Participation in another clinical study 28 days prior to dose.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
AUC0-t (area under the concentration-time curve) for entinostat administered with or without omeprazole (Part 1), with or without famotidine (Part 2), or omeprazole with and without acidic beverage | Pre-dose through Day 22
AUC0-inf (area under the concentration-time curve, from time 0 extrapolated to infinity for entinostat administered with or without omeprazole (Part 1), with or without famotidine (Part 2), or omeprazole with and without acidic beverage (Part 3) | Pre-dose through Day 22
Cmax (maximum observed concentration) for entinostat administered with or without omeprazole (Part 1), with or without famotidine (Part 2), or omeprazole with and without acidic beverage (Part 3) | Pre-dose through Day 22

SECONDARY OUTCOMES:
AUC%extrap (percent of AUC0-inf extrapolated) for entinostat administered with or without omeprazole (Part 1), with or without famotidine (Part 2), or omeprazole with and without acidic beverage (Part 3) | Pre-dose through Day 22
Tmax (time to reach maximum observed concentration) for entinostat administered with or without omeprazole (Part 1), with or without famotidine (Part 2), or omeprazole with and without acidic beverage (Part 3) | Pre-dose through Day 22
Kel (apparent terminal elimination rate constant) for entinostat administered with or without omeprazole (Part 1), with or without famotidine (Part 2), or omeprazole with and without acidic beverage (Part 3) | Pre-dose through Day 22

OTHER OUTCOMES:
T1/2 (apparent terminal elimination half-life) for entinostat administered with or without omeprazole (Part 1), with or without famotidine (Part 2), or omeprazole with and without acidic beverage (Part 3) | Pre-dose through Day 22
CL/F (apparent total plasma clearance after oral (extravascular) administration)for entinostat administered with or without omeprazole (Part 1), with or without famotidine (Part 2), or omeprazole with and without acidic beverage (Part 3) | Pre-dose through Day 22
Vz/F (apparent volume of distribution during the terminal elimination phase) for entinostat administered with or without omeprazole (Part 1), with or without famotidine (Part 2), or omeprazole with and without acidic beverage | Pre-dose through Day 22
Changes from baseline in physical exam | Baseline through Day 1
Changes from baseline in vital signs | Baseline through Day 22
Changes from baseline in ECG results | Baseline through follow Day 22
Changes from baseline in clinical laboratory tests | Baseline through Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sterling, MD, Principal Investigator — Celerion
Locations (2):
- United States (2):
  - Celerion, Tempe, Arizona
  - Celerion, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No
Data will be reviewed throughout the study by the sponsor, clinical research organization assisting with serious adverse event management, and routine monitoring to safeguard the interests of the trial subjects and to assess the safety of the interventions administered during the trial.